CLINICAL TRIAL: NCT04824521
Title: The Mindful Pregnancy Study: A Pilot Feasibility Study of Mindfulness-Oriented Recovery Enhancement With Pregnant Women With Opioid Use Disorder
Brief Title: A Pilot Feasibility Study of Mindfulness-Oriented Recovery Enhancement With Pregnant Women With Opioid Use Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol is determined to no longer be able to meet study objectives due to failure to enroll participants within the requisite time period.
Sponsor: University of Montana (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Sarah Reese, Assistant Professor of Social work, University of Montana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-21; 5P20GM130418 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-04-01 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Oriented Recovery Enhancement via tele-health (Experimental): Participants will be assigned to 8 weeks of Mindfulness-Oriented Recovery Enhancement delivered via tele-health.
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement — MORE is a mindfulness-based intervention.

SUMMARY:
Thirty pregnant women with substance use disorder will be recruited to participate in eight sessions of MORE.

DETAILED DESCRIPTION:
Participants will be asked to complete a battery of self-report measures and a semi-structured qualitative interview at three times points-before the intervention begins, after session four, and again after session eight. Participants will also be asked to complete self-report measures before and after each session. The primary aims of this study are as follows.

Aim 1: To adapt the in-person MORE intervention for telehealth delivery. Aim 2: To assess the overall feasibility and acceptability of this telehealth intervention. Hypothesis: MORE delivered via telehealth will be both feasible and acceptable to participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be pregnant.
* Must be able to communicate in English.
* Must have met criteria for opioid use disorder in the past year.

Exclusion Criteria:

* None.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Reese, Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began 2/10/21 upon IRB approval and ended on 5/1/22. Recruitment efforts included outreach to OBGYN providers, healthcare systems, pain management clinics, substance use treatment providers, community groups, and harm reduction services. Providers and community members were asked to refer potential participants to the study and to post flyers. The team also advertised online through social media.
Pre-assignment Details: We did not exclude any participants from the study before assignment to groups.
Period: Overall Study
Arm/Group | Mindfulness-Oriented Recovery Enhancement Via Tele-health
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness-Oriented Recovery Enhancement Via Tele-health
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 31 [31 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
SUD Symptoms - Mini Neuropsychiatric Interview - Alcohol Use Disorder [Mean (Full Range); unit: symptoms] — The Mini Neuropsychiatric Interview is a brief structured diagnostic interview for the major psychiatric disorders in the DSM-V. For this study, we conducted a structured interview with participants to determine the number of symptoms of substance use disorder they had experienced in the past year. After completing eight sessions of Mindfulness-Oriented Recovery Enhancement, we conducted the same interview to learn the number of symptoms of substance use disorder participants had experienced in the past eight weeks.
  symptoms | 12 [12 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction
Description: Participants will complete the Client Satisfaction Questionnaire.
Time Frame: 8 weeks
Population: Participant did not complete this measure.
Arm/Group | Mindfulness-Oriented Recovery Enhancement Via Tele-health
Number analyzed (Participants) | 0

2. Secondary Outcome: SUD Symptoms - Mini Neuropsychiatric Interview
Description: The Mini Neuropsychiatric Interview is a brief structured diagnostic interview for the major psychiatric disorders in the DSM-V. For this study, we conducted a structured interview with participants to determine the number of symptoms of substance use disorder they had experienced in the past year. After completing eight sessions of Mindfulness-Oriented Recovery Enhancement, we conducted the same interview to learn the number of symptoms of substance use disorder participants had experienced in the past eight weeks.
Time Frame: 8 weeks
Measure: Number; unit: symptoms
Arm/Group | Mindfulness-Oriented Recovery Enhancement Via Tele-health
Number analyzed (Participants) | 1
symptoms | 12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the time the participant was engaged in the study, about 10 weeks.
Arm/Group | Mindfulness-Oriented Recovery Enhancement Via Tele-health
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Unable to recruit the number of participants anticipated possibly due to stigma related to substance use in pregnancy, as well as challenges related to Covid-19 and the impact of the pandemic on healthcare and social service systems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04824521/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04824521/SAP_001.pdf